CLINICAL TRIAL: NCT00741013
Title: Imaging Biomarkers of Pulmonary Inflammation
Brief Title: Quantifying Airway Inflammation With Radiologic Tests
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-1137
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Lung Inflammation
Keywords: randomized; positron emission tomography; lung inflammation; lovastatin; recombinant human activated protein C; endotoxin; fluorodeoxyglucose
MeSH Terms: conditions — Pneumonia | interventions — Lovastatin; drotrecogin alfa activated; Endotoxins; Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo pill and placebo IV (Placebo Comparator)
  Interventions: Drug: placebo pill and placebo IV; Biological: Endotoxin
- Lovastatin pill and placebo IV (Experimental)
  Interventions: Drug: Lovastatin pill and placebo IV; Biological: Endotoxin
- Placebo pill and rhAPC IV (Experimental)
  Interventions: Drug: placebo pill and recombinant human activated protein C IV; Biological: Endotoxin

INTERVENTIONS:
Drug: placebo pill and placebo IV — Placebo pill every four hours, starting 16 hours before intrabronchial LPS and ending 24 hours after intrabronchial LPS
  Placebo IV starting 2 hours before intrabronchial LPS and ending 24 hours after intrabronchial LPS
  Arms: Placebo pill and placebo IV
Drug: Lovastatin pill and placebo IV — lovastatin pill every four hours, total of 80 milligrams a day, starting 16 hours before intrabronchial LPS and ending 24 hours after intrabronchial LPS
  Placebo IV starting 2 hours before intrabronchial LPS and ending 24 hours after intrabronchial LPS
  Other Names: Mevacor
  Arms: Lovastatin pill and placebo IV
Drug: placebo pill and recombinant human activated protein C IV — placebo pill every four hours, total of 80 milligrams a day, starting 16 hours before intrabronchial LPS and ending 24 hours after intrabronchial LPS
  recombinant human activated protein C IV 24 micrograms per kg per hour starting 2 hours before intrabronchial LPS and ending 24 hours after intrabronchial LPS
  Other Names: Xigris
  Arms: Placebo pill and rhAPC IV
Biological: Endotoxin — Endotoxin 4 ng/kg instilled bronchoscopically in all volunteers 12 hours after starting lovastatin treatment and 2 hours after starting recombinant human activated protein C treatment.
  Other Names: Reference Endotoxin (E. Coli O113:H10K); lipopolysaccharide

SUMMARY:
In this randomized, double-blind, placebo controlled trial we used positron emission tomography to determine if lovastatin or recombinant human activated protein C exhibit anti-inflammatory effects in humans following intrabronchial installation of lipopolysaccharide (LPS or endotoxin).

DETAILED DESCRIPTION:
Quantitative, noninvasive biomarkers for lung-specific inflammation have yet to be developed but can potentially contribute significantly to the development of therapies to treat lung inflammation. The purpose of this study was to demonstrate that positron emission tomographic (PET) imaging with [18F}fluorodeoxyglucose (FDG-PET) can be used to quantify the change in lung inflammation in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, man or woman, any race or ethnicity, age 19 - 44 years old
* Screening FEV1 and FVC must be > 80% of predicted.
* Screening oxygen saturation by pulse oximetry is >97% on room air.
* Research volunteer must be capable of lying still and supine within the PET scanner for ~2 ½ hours.
* Research volunteer must be capable of fasting for 6 hours.

Exclusion Criteria:

* Pregnancy (confirmed by a qualitative urine hCG pregnancy test)
* Lactation.
* Actively menstruating at time of randomization
* History of tobacco use or has smoked other illicit drugs (marijuana, cocaine) in the past year.
* Research volunteer is currently taking any prescription medications.
* Research volunteer is at increased risk for radiation exposure (e.g. flight attendants)
* Research volunteer is enrolled in another research study of an investigational drug.
* Research volunteer has a known allergy to both trimethoprim/sulfamethoxazole and amoxicillin.
* Research volunteer has a known allergy to drugs routinely used during bronchoscopy.
* Research volunteer has a known allergy to lovastatin or rhAPC
* Fasting glucose at time of PET study > 150 mg/dl.
* Exclusion criteria related to use of rhAPC:

  * Active or history of internal bleeding within the past 3 months
  * History of hemorrhagic stroke within the past 3 months.
  * History of intracranial or intraspinal surgery, or severe head trauma, within the past 3 months
  * History of trauma with an increased risk of life-threatening bleeding within the past 3 months
  * History of receiving thrombolytic therapy within the past 3 months.
  * History of receiving oral anticoagulants or glycoprotein IIb/IIIa inhibitors within the past 3 months.
  * History of using aspirin > 650 mg/d or other platelet inhibitors within the past 7 days.
  * Any history of intracranial arteriovenous malformation or aneurysm
  * Any history of a known bleeding diathesis
  * Any history of chronic severe hepatic disease
  * Presence of an epidural catheter
  * Any history of intracranial neoplasm or mass lesion or evidence of cerebral herniation
  * Use of heparin during past 7 days
  * Platelet count <100,000 x 106/L
  * Prothrombin time-INR > 1.5
  * SGOT >47 IU/L, SGPT > 53 IU/L, or bilirubin > 1.1 mg/dl
  * Any other condition in which bleeding constitutes a significant hazard or would be particularly difficult to manage because of its location.
* Exclusion criteria related to use of lovastatin:

  * History of chronic active liver disease or acute liver disease within the past 3 months
  * SGOT >47 IU/L, SGPT > 53 IU/L, or bilirubin > 1.1 mg/dl.

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Delphine L Chen, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Chen DL, Bedient TJ, Kozlowski J, Rosenbluth DB, Isakow W, Ferkol TW, Thomas B, Mintun MA, Schuster DP, Walter MJ. [18F]fluorodeoxyglucose positron emission tomography for lung antiinflammatory response evaluation. Am J Respir Crit Care Med. 2009 Sep 15;180(6):533-9. doi: 10.1164/rccm.200904-0501OC. Epub 2009 Jul 2. PMID 19574441

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Pill and Intravenous (i.v.) Placebo: Control group receiving only placebo drug interventions
- Lovastatin Pill and i.v. Placebo: Group receiving lovastatin as the primary drug intervention
- Placebo Pill and Recombinant Human Activated Protein C i.v.: Group receiving recombinant human activated protein C (rhAPC) as the drug intervention
Period: Overall Study
Arm/Group | Placebo Pill and Intravenous (i.v.) Placebo | Lovastatin Pill and i.v. Placebo | Placebo Pill and Recombinant Human Activated Protein C i.v.
Started | 7 | 8 | 7
Completed | 6 | 6 | 6
Not Completed | 1 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Discovered failed screen after enrolled | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Pill and Intravenous (i.v.) Placebo | Lovastatin Pill and i.v. Placebo | Placebo Pill and Recombinant Human Activated Protein C i.v. | Total
Number analyzed (Participants) | 7 | 8 | 7 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 7 | 22
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 5 | 6 | 6 | 17
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Ki (Measure of [18F]Fluorodeoxyglucose ([18F]FDG) Uptake Determined by Patlak Graphical Analysis) in the Right Lung 24 Hours After LPS Instillation
Description: Calculated Ki was used to measure the amount of lung inflammation before and after instillation of endotoxin to assess the effect of placebo, lovastatin, and rhAPC treatment
Time Frame: 24 hours after endotoxin instillation
Measure: Mean (Standard Deviation); unit: Change in Ki
Arm/Group | Placebo Pill and Intravenous (i.v.) Placebo | Lovastatin Pill and i.v. Placebo | Placebo Pill and Recombinant Human Activated Protein C i.v.
Number analyzed (Participants) | 6 | 6 | 6
Change in Ki | 18.8 (9.2) | 8.4 (4.3) | 14.2 (7.4)
Statistical Analysis 1: Comparison: Placebo Pill and Intravenous (i.v.) Placebo vs Lovastatin Pill and i.v. Placebo vs Placebo Pill and Recombinant Human Activated Protein C i.v; One-way analysis of variance was performed to determine whether lovastatin or rhAPC effectively reduced endotoxin-induced lung inflammation; Test type: Superiority or Other; p < 0.05, ANOVA — Only a single statistical analysis was performed upon completion of the study

2. Secondary Outcome: Number of Total Nucleated Cells From Bronchoalveolar Lavage (BAL) Fluid 24 Hours After Endotoxin Instillation
Description: Number of total nucleated cells isolated from the first aliquoe of BAL obtained to correlate with PET data.
Time Frame: 24 hours after endotoxin instillation
Measure: Mean (Standard Deviation); unit: cells per cubic mm
Arm/Group | Placebo Pill and Intravenous (i.v.) Placebo | Lovastatin Pill and i.v. Placebo | Placebo Pill and Recombinant Human Activated Protein C i.v.
Number analyzed (Participants) | 6 | 6 | 6
cells per cubic mm | 545 (425) | 311 (237) | 520 (196)

ADVERSE EVENTS:
Arm/Group | Placebo Pill and Intravenous (i.v.) Placebo | Lovastatin Pill and i.v. Placebo | Placebo Pill and Recombinant Human Activated Protein C i.v.
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 5/8 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Pill and Intravenous (i.v.) Placebo (N=7) | Lovastatin Pill and i.v. Placebo (N=8) | Placebo Pill and Recombinant Human Activated Protein C i.v. (N=7)
Decreased pulmonary function (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — A drop of greater than 20% from baseline in FEV1 was considered a serious adverse event warranting withdrawal from the study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Pill and Intravenous (i.v.) Placebo (N=7) | Lovastatin Pill and i.v. Placebo (N=8) | Placebo Pill and Recombinant Human Activated Protein C i.v. (N=7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) — Symptom reported within 48 hours of endotoxin administration.
Fever (General disorders) | 3 (4) | 2 (2) | 2 (2)
Headache (General disorders) | 2 (2) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash under neck (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Body ache (General disorders) | 1 (1) | 1 (1) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
General body discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No